CLINICAL TRIAL: NCT01088867
Title: Using DNIC to Predict Acupuncture Therapy Outcome: A Pilot Study
Brief Title: Using Diffuse Noxious Inhibitory Control (DNIC) to Predict Acupuncture Therapy Outcome: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Bastyr University (Other)
Responsible Party: Principal Investigator, Ruth Landau, Professor, Director of OB Anesthesia & Clinical Genetics Research, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 36255-A
Record Dates: First submitted 2010-03-12; First posted 2010-03-17 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Pain
Keywords: Pain; Acupuncture; DNIC; Electroacupuncture
MeSH Terms: conditions — Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acupuncture (Other): 14 weeks of electroacupuncture therapy.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Electroacupuncture
  Other Names: Pantheon Electroacupuncture Device

SUMMARY:
The investigators hypothesize that acupuncture modifies the DNIC efficiency and that DNIC can serve as a predictor to identify 'good responders' to acupuncture early in therapy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women with a progesterone-coated intrauterine device (Mirena), and
* Men greater than or equal to 18 years old.

Exclusion Criteria:

* Acupuncture treatment in the previous six weeks, to discount any persisting effect of acupuncture.
* Treatment of a pain condition with pain medication.
* Regular use of benzodiazepines.
* Skin diseases, such as scleroderma, psoriasis or eczema.
* An adverse event due to acupuncture therapy.
* Pregnant women.
* Women without a progesterone-coated intrauterine device (Mirena).
* Anyone older than 60 years of age, fatigued, with a pacemaker ICD, artificial joint, prolonged bleeding time/hemophilia, open wounds, or a known susceptibility to profound analgesia after acupuncture treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Diffuse Noxious Inhibitory Control Efficiency | Week 0, 2, 4, 6, and 12 of acupuncture therapy
  The efficiency of diffuse noxious inhibitory control (DNIC) is a measure of one's ability to inhibit pain perception. DNIC efficiency is assessed by a psychophysical test that involves a heat thermode as the "test stimulus" and a warm water bath as the "conditioning stimulus". The results of this test will be used as the primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Landau, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States